CLINICAL TRIAL: NCT01876680
Title: The Effects (Pain, Function, Biochemistry and Psychological Factors) of Two Different Home-exercise Programmes on Women Suffering Long Term Nack/Shoulder Muscle Pain
Brief Title: The Effects of Two Different Home-exercise Programmes on Women Suffering Long Term Neck/Shoulder Muscle Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Bjorn Gerdle, Professor MD, Rehabilitation Medicine, Linkoeping University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LIU-001
Record Dates: First submitted 2011-09-05; First posted 2013-06-12 (Estimated); Last update posted 2013-06-12 (Estimated); Status verified 2013-06

CONDITIONS: Neck Pain
Keywords: chronic; neck; shoulder; exercise
MeSH Terms: conditions — Neck Pain; Bronchiolitis Obliterans Syndrome; Motor Activity | interventions — Exercise; Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1: Stretching and aerobic exercise (Experimental): Group 1 undertook a stretching programme for neck/shoulder muscles three times weekly and performed aerobic exercise för 30 minutes three times weekly.
  Interventions: Other: Stretching and aerobic exercise
- Group 2: Strength training (Experimental): Group 2 undertook a stretching programme for neck/shoulder muscles three times weekly, performed aerobic exercise three times weekly and performed weight training using dumbbells for the neck/shoulder area and exercises to strengthen core and leg muscles for 45 minutes three times weekly.
  Interventions: Other: Strength training

INTERVENTIONS:
Other: Stretching and aerobic exercise — Stretching programme for neck/shoulder muscles three times weekly and aerobic exercise för 30 minutes three times weekly.
  Participants kept exercise diaries and physiotherapist provided support over the phone or through e-mail. The intervention lasted one year.
  Arms: Group 1: Stretching and aerobic exercise
Other: Strength training — Stretching programme for neck/shoulder muscles three times weekly, aerobic exercise för 30 minutes three times weekly and weight training using dumbbells for the neck/shoulder area and exercises to strengthen core and leg muscles for 45 minutes three times weekly.
  Participants kept exercise diaries and physiotherapist provided support over the phone or through e-mail. The intervention lasted one year.
  Arms: Group 2: Strength training

SUMMARY:
The purpose of this study is to investigate the effects of specific neck/shoulder muscle exercises on pain, function, biochemistry and psychological factors in women suffering chronic neck/shoulder pain.

ELIGIBILITY:
Inclusion Criteria:

* female
* 20-60
* long term neck/shoulder muscle pain
* willing to exercise

Exclusion Criteria:

* widespread pain
* pregnancy
* major trauma in medical history
* tendonitis in upper extremities
* neurological causes of the pain
* inflammatory and hormonal disorders

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2009-09; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Pain | Before training, 4-6 months and after one year of training.
  Methods of measurement: Surveys, physical tests, microdialysis.
Function | Before training, 4-6 months and after one year of training.
  Methods of measurement: Surveys, physical tests, microdialysis.

SECONDARY OUTCOMES:
Muscle biochemistry | Before training, 4-6 months follow-up and 12 months follow-up
  Biochemical substances from the interstitium of the trapezius muscle will be determined eg, serotonin, glutmate, lactate, pyruvate, endocannabinoids.
Psychological factors | Before training, 4-6 months follow-up and 12 months follow-up
  Aspects concerning psychological distress will be followed eg depression and anxiety using Hospital Anxiety and Depression Scale (HADS).
Pain sensitivity | Before training, 4-6 months follow-up and 12 months follow-up
  Pain thresholds for pressure (algometry) and heat and cold (QST) will be registered.

CONTACTS AND LOCATIONS:
Overall Officials: Britt Larsson, Assoc Prof, Principal Investigator — rehabilitation medicine, Faculty of Health Sciences, Linköping University, SE 581 85, Linköping, Sweden
Locations (1):
- Faculty of Health Sciences, Linköping University, Linköping, Östergötland County, Sweden

REFERENCES:
- [Derived] Ghafouri N, Ghafouri B, Fowler CJ, Larsson B, Turkina MV, Karlsson L, Gerdle B. Effects of two different specific neck exercise interventions on palmitoylethanolamide and stearoylethanolamide concentrations in the interstitium of the trapezius muscle in women with chronic neck shoulder pain. Pain Med. 2014 Aug;15(8):1379-89. doi: 10.1111/pme.12486. Epub 2014 Jul 4. PMID 24995488
- [Derived] Karlsson L, Takala EP, Gerdle B, Larsson B. Evaluation of pain and function after two home exercise programs in a clinical trial on women with chronic neck pain - with special emphasises on completers and responders. BMC Musculoskelet Disord. 2014 Jan 8;15:6. doi: 10.1186/1471-2474-15-6. PMID 24400934
- See also: Related Info — http://www.liu.se